CLINICAL TRIAL: NCT07308886
Title: Phase II Study of Recombinant Glycosylated Human Interleukin-7 (CYT107) for the Treatment of Kaposi Sarcoma in Participants With HIV and Immune Non-response (REGIMEN-KS HIV)
Brief Title: Recombinant Glycosylated Human Interleukin-7 (CYT107) for the Treatment of Kaposi Sarcoma in Participants With HIV and Immune Non-Response (REGIMENKS HIV)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002361; 002361-C
Record Dates: First submitted 2025-12-24; First posted 2025-12-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Kaposi Sarcoma
Keywords: human herpesvirus 8; KS-associated herpes virus; HIV; Interleukin-7; Lymphoproliferative Disorder
MeSH Terms: conditions — Sarcoma, Kaposi; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Treatment with CYT107
  Interventions: Drug: CYT107

INTERVENTIONS:
Drug: CYT107 — CYT107 is administered by IM injections at 20 mcg/kg every week for up to 4 weeks/4 doses

SUMMARY:
Background:

Kaposi sarcoma (KS) is a cancer that causes abnormal tissue to grow in the skin, lymph nodes, and other organs. KS is caused by a virus known as Kaposi sarcoma herpesvirus. People infected with human immunodeficiency virus (HIV) account for 80% of KS cases in the United States. Having HIV can weaken the immune system and this can lead to KS. Weaker immune systems may be measured by low T cells (a type of immune cell). CYT107 is a human protein, made in a laboratory, that may help boost immunity, specifically by increasing T cells, in people with HIV-associated KS.

Objective:

To see if CYT107 can shrink KS tumors.

Eligibility:

People aged 18 years and older with HIV-associated KS.

Design:

Participants will be screened. They will have a physical exam with blood tests. Their skin lesions will be measured. They will have an x-ray of their lungs. Their ability to perform everyday tasks will be reviewed. A sample of lesion tissue (biopsy) may be collected from the skin.

CYT107 is injected into the muscle of the arm, buttocks, or lower thigh once a week for up to 4 weeks. Participants will receive the shots at the clinic. Blood and other tests will be repeated at each visit. KS lesions will be measured and photographed on the 1st and 4th visits.

Participants who improved after the first 4 weeks may have another 4-week treatment within a year.

Follow-up visits will continue for 3 years.

DETAILED DESCRIPTION:
Background:

* Kaposi sarcoma (KS) is an angioproliferative tumor associated with KS-associated herpes virus (KSHV), also known as human herpesvirus 8 or (HHV-8) infection.
* Human immunodeficiency virus (HIV) infection-related KS accounts for greater than 80% of KS in the United States.
* Survival rates from HIV-related KS are poorer than classic KS, despite improving substantially with the introduction of antiretroviral therapy (ART).
* KS oncogenesis is associated with loss of T-cell mediated control of KSHV, the viral cause of KS.
* While treatment of persons with HIV (PWH) with ART can improve T-cell counts and immunity, their T-cell counts often do not return to normal and they are often left with residual immunodeficiency.
* There are a group of patients who have well controlled HIV but continue to have low CD4 T-cell counts (<=350 cells/mcL) who are termed immune non-responders . This group possess a high rate of KS persistence, and chemotherapy can often contribute to

lymphopenia.

* The cytokine interleukin-7 (IL-7) plays an important role in T-cell development and proliferation and regulates T-cell homeostasis throughout life.
* IL-7 administration is very potent at producing new T cells such as na(SqrRoot) ve T cells and recent thymic emigrants.
* Administration of short acting recombinant human IL-7 was well-tolerated and has resulted in a dose-dependent increase in peripheral T cells and broadening of T-cell receptor (TCR) diversity.

Objective:

-To assess the overall response rate (ORR) of CYT107 defined as the best response (complete response [CR], clinical complete response [CRR], partial response [PR]) within 24 weeks in the first course of treatment, using the modified AIDS Clinical Trial Group

(ACTG) KS response criteria in immune non-response participants with HIV-associated KS who had prior systemic KS therapy or who are KS therapy naive

Eligibility:

* Age >=18 years
* Histologically confirmed diagnosis of KS in people with HIV.
* All participants should have at least five (5) measurable cutaneous KS lesions.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <=3
* CD4 T cell count <=350 cells/mcL
* This is an open label, nonrandomized Phase II study assessing the safety and activity of CYT107 in participants with HIV-associated KS.
* Participants will be enrolled in two cohorts based on prior exposure to KS therapy.
* A safety run-in will be conducted for the first 12 participants with no more than three participants treated simultaneously.
* Participants will receive CYT107 at 20 mcg/kg by intramuscular (IM) injections every week for up to 4 weeks/4 doses.
* Participants who have an increase in CD4 T-cell count following administration of CYT107 and evidence of KS response per ACTG criteria but subsequently experience a decrease in CD4 T-cell count (>=100 cells/mcL) with associated deterioration in KS, or have

had prior systemic KS therapy and first course resulted in SD only, may be eligible to receive a second course of CYT107 administration (for up to 4 weeks/4 doses).

-Up to 29 evaluable participants will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA
* Histologically confirmed KS by NCI Laboratory of Pathology (LP), with or without any prior systemic KS treatment
* Participants with HIV infection
* Age >= 18 years
* All participants should have at least five (5) measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion.
* Participants with stage T1 KS with visceral involvement must:

  * have any/all associated tumor associated symptoms <= Grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 criteria and/or,
  * require no immediate intervention (e.g., mild oozing of oral KS is allowed).
* Participants did not receive prior systemic therapy for KS or received prior systemic therapy and currently are either plateau in response, relapsed disease, progressive disease (PD), or inadequate response to treatment. Note: Previous local therapy or radiation is not considered systemic therapy.
* Participants must:

  * have been on effective ART therapy for at least 2 months prior to the study drug initiation and
  * have HIV VL <= 100 copies/mL and
  * have persistent KS, affecting quality of life due to either T1 or T0 disease with inadequate disease regression on ART alone.
* ECOG PS <=3
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count (ANC) >= 500/mcL
  * platelets >= 50,000/mcL
  * hemoglobin (hgb) >= 8g/dL
  * total bilirubin <= 1.5 institutional upper limit of normal (iULN) or <3 x iULN for Gilbert s syndrome or HIV protease inhibitors
* AST <= 2.5 x iULN
* ALT <= 2.5 x iULN
* CD4 T-cell count <= 350/mcL
* Participants must be willing to co-enroll to protocol 17C0174 "Molecular Characterization of Viral-associated Tumors, Tumors occurring in the Setting of HIV or other Immune Disorders and Castleman Disease"
* Participants with chronic hepatitis B virus (HBV) infection are eligible if they are on suppressive antiviral therapy.
* Participants with a hepatitis C virus (HCV) infection must have an undetectable HCV VL due to prior treatment or natural resolution.
* Women of child-bearing potential (WOCBP) and men able to father a child must agree to use an effective method of contraception (hormonal, barrier, surgical sterilization, abstinence) at the study entry, for the duration of study therapy, and for up to 4 months

after discontinuation of study drug.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 4 months after the last dose of the study drug.
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA

-Participants who have not recovered from immune-related AEs due to prior therapy (i.e., have residual toxicities > Grade 1 per CTCAE v.5.0).

Note: Participants with hypothyroidism managed by supplemental levothyroxine are eligible.

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to Chinese Hamster Ovary (CHO) cell products, chimeric or humanized antibodies or fusion proteins.
* Participants must not have received chemotherapy, radiotherapy, or other KS directed therapy other than ART for HIV within 2 weeks before the initiation of study drug.
* Participants must not have received treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents) or systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or IL-2, pomalidomide, or immune checkpoint inhibitors) within 2 weeks before initiation of study treatment.

Note: Participants who have received acute, low dose of systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled. The use of inhaled corticosteroids, and mineralocorticoids (e.g., fludrocortisone) for participants with orthostatic hypotension or adrenocortical insufficiency is allowed.

* History or risk of autoimmune disease, except for:

  * the presence of laboratory evidence of autoimmune disease (e.g., history of positive antinuclear antibody [ANA] titer or lupus anticoagulant) without associated symptoms,
  * clinical evidence of vitiligo or other forms of depigmenting illness; and/or,
  * mild autoimmunity not impacting the function of major organs (e.g., limited psoriasis).
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (e.g., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest x-ray.

Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

* History of allogeneic stem cell transplant and all other organ transplant.
* Another prior or concurrent malignancy requiring active therapy
* Active tuberculosis
* Positive serum or urine beta-human chorionic gonadotropin (beta-hCG) test at screening.
* Participants must not have received prohibited therapies within 4 weeks before initiation of study treatment
* Severe uncontrolled intercurrent illness that would limit compliance with study requirements, as evaluated by history, physical exam, and chemistry panel.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2036-01-31 (Estimated); Study Completion 2037-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit | Baseline/prior to treatment (week 1/cycle 1), at cycle 4 (week 4), at EOT (week 8), at safety visits (weeks 12 and 16), and in follow-up (week 24 )
  Percentage of participants with the best overall response of CR, CRR, or PR to therapy.

SECONDARY OUTCOMES:
Safety of CYT107 | Prior to each cycle, at EOT (week 8), and at safety visits (weeks 12 and 16)
  Adverse events (AEs) will be reported by type and grade of toxicity
Time of duration of response | Baseline/prior to treatment (week 1/cycle 1), at cycle 4 (week 4), at EOT (week 8), at safety visits (weeks 12 and 16), and in follow-up (up to 3 years post-treatment)
  The interval between initiating therapy and the time to disease progression in patients who achieve CR, PR, or SD.
Time of progression free survival | Baseline/prior to treatment (week 1/cycle 1), at cycle 4 (week 4), at EOT (week 8), at safety visits (weeks 12 and 16), and in follow-up (up to 3 years post-treatment)
  The interval between initiating therapy and the time to disease progression or death, whichever happens first
Proportion of participants requiring a second course of CYT107. | ongoing
  Percentage of participants who meet criteria and receive second course of treatment
Clinical benefit of a second course of CYT107 | Baseline/prior to treatment (week 1/cycle 1), at cycle 4 (week 4), at EOT (week 8), at safety visits (weeks 12 and 16), and in follow-up (week 24 )
  Percentage of participants that received a second course with the best overall response of CR, CRR, or PR to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002361-C.html